CLINICAL TRIAL: NCT03829865
Title: Chicago Classification Normative Metrics in a Healthy Russian Cohort According to High-resolution Esophageal Manometry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vasily Isakov, MD, PhD, Professor, AGAF, Russian Academy of Medical Sciences
Other Study IDs: OGIG-2019-1
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Water-perfused HREM: Healthy volunteers examined with water-perfused high resolution esophageal manometry
  Interventions: Diagnostic Test: High resolution esophageal manometry
- Solid-state HREM: Healthy volunteers examined with high resolution esophageal manometry with solid-state catheter
  Interventions: Diagnostic Test: High resolution esophageal manometry

INTERVENTIONS:
Diagnostic Test: High resolution esophageal manometry — High resolution esophageal manometry will be performed to eligible subjects willing to participate in the study

SUMMARY:
High resolution esophageal manometry normative values are still need to be studied in different populations and with the use of solid-state and water-perfused systems. There has been no study on the subject in healthy Russian population yet.

DETAILED DESCRIPTION:
High-resolution esophageal manometry (HREM) is the current modality used to evaluate esophageal motility. There are 2 types of system: water-perfused system that is cheaper to maintain and a solid-state system that is considered to be more sensitive. According to the data obtained in the study of 400 patients and 75 controls by J Pandolfino et al it was proposed to use a common algorithm of HREM data interpretation and the normative values of the parameters used to interpret the color plots of HREM. This formed the basis for the first version of the currently used HREM reporting algorithm and classification of esophageal motility disorders called Chicago Classification (CC). To date, this classification has been updated several times by the International Working Group based on the recently published data. The Working group stated that the proposed normative values still need to be widely studied for each HREM system and in different populations. Some studies has been published recently on the normative values of HREM in different countries (predominantly in the US, in some European countries, Korea, India and China. But there has been no study on the subject in Russia still.

ELIGIBILITY:
Inclusion Criteria (all points are necessary for inclusion):

* Willingness to participate on the basis of signed informed consent form;
* Patients of both sexes, aged 18 to 65 years inclusive;
* Permanent residence in the Russian Federation;
* Absence of esophageal diseases, confirmed by the results of clinical and instrumental examination
* Ability to follow instructions during high-resolution esophageal manometry procedure

Exclusion Criteria (patient is not eligible when at least one exclusion criterion is met):

* diseases of the esophagus (any condition on the basis of clinical and / or instrumental examination, including: complaints of heartburn, belching, difficulty to swallow solid and/or liquid food;
* any surgical intervention on the gastrointestinal tract and / or chest organs in medical history;
* solid organ transplantation in medical history with the exception of a corneal transplant and surgery to replace the lens of the eye;
* any oncology of any localization except for skin cancer in situ in the medical history;
* any decompensated diseases of any organs and systems, which, in the opinion of the researcher, makes it impossible to carry out the procedure of esophageal manometry of high resolution or if the procedure may cause the risk of deterioration of the patient's condition;
* any condition, clinical and laboratory signs of alcohol abuse (abuse will be assessed in the case of male subjects consuming more than 30 g of pure alcohol per day and using more than 20 g of pure alcohol per day by female subjects;
* any illegal drug use, current or past;
* use of concomitant medications that can affect esophageal motility including, but not limited to: calcium channel blockers, metoclopramide, m-cholinolytics, domperidone, erythromycin, nitrates, tricyclic antidepressants, opiates, beta-blockers, beta-adrenomimetics, alcohol. The duration of the period of non-use of these drugs should provide sufficient time for the complete cessation of their pharmacological action, but not less than two half-life.
* pregnant or breastfeeding women
* any condition making impossible to perform high resolution esophageal manometry (previously known poor tolerability of the procedure; narrow nasal passages; significant curvature of the nasal septum etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is aimed to evaluate high resolution esophageal motility parameters in subjects who have no signs of any esophageal disorders and are residents of Russia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean IRP | mean value of 10 swallows by 30 seconds (about 7 minutes per subject)
  Integrated Relaxation Pressure - mean of the 4 s of maximal deglutitive relaxation in the 10-s window beginning at upper esophageal sphincter relaxation
Mean DCI | mean value of 10 swallows by 30 seconds (about 7 minutes per subject)
  distal contractile integral - Amplitude x duration x length (mmHg x s x cm) of the distal esophageal contraction exceeding 20 mmHg from the transition zone to the proximal margin of the LES
Mean DL | mean value of 10 swallows by 30 seconds (about 7 minutes per subject)
  distal latency - Interval between UES relaxation and the contractile deceleration point
Mean upper esophageal sphincter mean resting pressure | mean value based on 30 seconds measurement of a subject
  mean pressure of the upper esophageal sphincter
Mean lower esophageal sphincter mean resting pressure | mean value based on 30 seconds measurement of a subject
  mean pressure of the upper esophageal sphincter

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, MD, PhD, Study Chair — Federal Research Center of Nutrition and Biotechnology; Sergey Morozov, MD, PhD, Principal Investigator — Federal Research Center of Nutrition and Biotechnology
Locations (3):
- Russia (3):
  - Gastroenterology and Hepatology, FRC Nutrition and Biotechnology, Moscow
  - Moscow clinical hospital #31, Moscow
  - Pavlov First Saint Petersburg State Medical University. Endoscopy Department, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Depersonalized individual data may be shared upon the study completion.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years
Access Criteria: by request